CLINICAL TRIAL: NCT05373940
Title: Cardioverter DefIbriIlator PlacEMent for priMary Prevention of Sudden cArdiac Death in Patients Older Than 70 Years: A Randomized Controlled Trial
Brief Title: Cardioverter DefIbriIlator PlacEMent for priMary Prevention of Sudden cArdiac Death in Patients Older Than 70 Years
Acronym: DILEMMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APHP200035; 2021-A01959-32 (Other: IDRCB)
Record Dates: First submitted 2022-04-20; First posted 2022-05-13 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure; Primary Prevention of Sudden Cardiac Death; Implantable Cardioverter Defibrillator
Keywords: Heart Failure; Prevention strategy of Sudden Cardiac Death; Implantable cardioverter defibrillator; Heart Failure Optimal Therapy; Mortality
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: This is a 2-arm parallel non-inferiority, randomized, open label, multicenter trial.
Who Masked: Outcomes Assessor
Masking Description: Three experts in cardiac electrophysiology and ICD will be in charge of uniformly approving, while blinded to the study group, ICD tracings, cardiovascular events, including specific causes of death, in order to validate the primary and secondary endpoints.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart failure optimal therapy alone (HFOT) (Experimental): Heart failure Optimal therapy without implantable cardioverter defibrillator. This group will not undergo an ICD implantation. They will be treated according to the HFOT recommended in the latest guidelines.
  Interventions: Device: No ICD implantation
- Heart failure optimal therapy (HFOT) + Implantable cardioverter defibrillator (ICD) (Active Comparator): Optimal medical therapy + implantable cardioverter defibrillator (HFOT+ICD). This group will undergo an ICD implantation (standard of care), any brand, CE marked, implantable (lifelong), available and reimbursed in the French market (the type and manufacturer at the discretion of the local investigator) in addition to heart failure medical therapy optimization.
  Interventions: Device: ICD implantation

INTERVENTIONS:
Device: ICD implantation — This group will undergo an ICD implantation (type and manufacturer at the discretion of the local investigator) in addition to heart failure medical therapy optimization.
  Patients of the "HFOT+ICD" group will be scheduled for ICD implantation.
  Arms: Heart failure optimal therapy (HFOT) + Implantable cardioverter defibrillator (ICD)
Device: No ICD implantation — Patients of the "HFOT alone" group will not undergo ICD implantation (except if they develop sustained ventricular arrhythmias and fulfil for secondary prevention ICD implantation), and continue with medical therapy optimization only.
  Arms: Heart failure optimal therapy alone (HFOT)

SUMMARY:
The primary objective of DILEMMA study is to assess whether the "heart failure optimal therapy alone (HFOT)" strategy is non inferior to the "HFOT+ICD" strategy in terms of overall survival 48 months after randomization, in patients ≥ 70 years with an ICD indication for primary prevention of SCD whether there is an indication for cardiac resynchronization therapy or not.

DETAILED DESCRIPTION:
Rationale Although not recognized by guidelines, there is no available data demonstrating the benefit of Implantable Cardioverter Defibrillator (ICD) for primary prevention strategy of Sudden Cardiac Death (SCD) in elderly. Nevertheless, ICD are currently implanted in this population by extending the results obtained in randomized trials involving younger subjects to the elderly. Finally, if the absence of implantation in the elderly was not inferior to the implantation of such a device, the non-implantation would avoid the device-related complications and decrease the health costs.

Main objective The primary objective of DILEMMA study is to assess whether the "heart failure optimal therapy alone (HFOT)" strategy is non inferior to the "HFOT+ICD" strategy in terms of overall survival 48 months after randomization, in patients ≥ 70 years with an ICD indication for primary prevention of SCD whether there is an indication for cardiac resynchronization therapy or not.

Design This is a 2-arm parallel non-inferiority, randomized, open label, multicenter trial. 730 patients will be included over 4 years. Follow up will last 4 years.

ELIGIBILITY:
Inclusion Criteria:

* ≥70 years old,
* Left ventricular ejection fraction ≤ 35%
* NYHA class II or III
* Heart failure HFOT ≥ 3 months
* Providing informed consent
* Affiliated to a French Health Insurance system.

Exclusion Criteria:

* Enrolled in or planning to enroll in a conflicting interventional trial
* Prior unstable sustained ventricular arrhythmia requiring external cardioversion
* Myocardial infarction within the 40 days
* Coronary artery intervention (catheter or surgical) within 90 days
* History of syncope in the previous 6 months
* Advanced cerebrovascular disease
* Cognitive impairment leading to the incapacity of consent
* Any disease other than cardiac disease (e.g. cancer, uremia, liver failure), associated with a likelihood of survival less than 1 year.
* Patient under tutorship, curatorship, or legal safeguard
* Persons deprived of their liberty by judicial or administrative decision (prisoner)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 730 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 48 months after randomization
  The primary endpoint will be the overall survival at 48 months after randomization to "HFOT alone" group or "HFOT+ICD" group.
  There is an annual follow-up with precise date of the fatal event and specific cause of death adjudicated by the blinded event committee.

SECONDARY OUTCOMES:
Cardiovascular mortality | 48 months after randomization
  Rate of cardiovascular mortality assessed by a blinded endpoint committee.
Sudden cardiac death and death from ventricular arrhythmias | 48 months after randomization
  Rate of sudden cardiac death and rate of death from ventricular arrhythmias assessed by a blinded endpoint committee.
Unplanned hospitalization due to cardiovascular causes | 48 months after randomization
  Number of unplanned hospitalization due to cardiovascular causes
ICD related complications including inappropriate therapies | 48 months after randomization
  Number of ICD related therapies (antitachycardia pacing and shocks), hematoma, infection related to the device, lead dislodgement requiring intervention, pneumothorax and tamponade.
Global quality of life score with 36-Item Short Form Survey (SF36) | baseline, 6, 12, 24, 36 and 48 months
  Global quality of life score with SF36 (Short form 36 health survey) : the norm data is 0-100, the health related quality of life is increased as the scores are increased.
Health-related quality of life score Euroqol EQ-5D questionnaire | baseline, 6, 12, 24, 36 and 48 months
  Health-related quality of life measured by using the European Quality Of Life (EQ-5D) auto-questionnaire. The digits for the five dimensions are combined into a 5-digit number that describes the patient's health state. The visual analogue scale (VAS) records the patient's self-rated health on a vertical axis from 0 (worst health) to 100 (best health)
Patient's global self-assessment of heart failure-related quality of life score | baseline, 6, 12, 24, 36 and 48 months
  The Minnesota Living with Heart Failure will be used to measure the subjects perception of how their heart failure affect their life. Norm data is 0-105 (21 items ; score 0-5), quality of life increases as scores decrease.
The Incremental cost-utility ratio. (ICUR) | 48 months
  The ICUR is calculated by dividing the difference between the average costs of both groups by the difference in mean QALYs gained in both groups. The QALYs will be constructed with the EuroQoL-5D (EQ-5D) questionnaire and value sets.
The incremental cost-effectiveness ratio (ICER) | 48 months
  The ICER will estimate the cost per additional survivor and is calculated by dividing the difference between the average costs of both groups by the difference in effectiveness (survival) between both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Eloi MARIJON, MD, PhD, Principal Investigator — AP-HP, Hôpital européen Georges Pompidou, Paris; Rodrigue GARCIA, MD, PhD, Study Director — CHU Poitiers, France
Locations (19):
- France (19):
  - Centre Hospitalier d'Aix en provence, Aix-en-Provence
  - CHU Amiens-Picardie-Site sud, Amiens
  - HôpitalHenri Mondor, Créteil
  - CHU Grenoble Alpes, La Tronche
  - Groupement d'Hôpitaux de l'Institut Catholique de Lille, Lomme
  - Hôpital de La Timone, Marseille
  - Hôpital de Brabois, Nancy
  - CHU de Nantes, Nantes
  - Hôpital Privé du Confluent, Nantes
  - Hôpital européen Georges Pompidou, Paris
  - Hôpital Pitié-Salpétrière, Paris
  - Hôpital Bichat - Claude Bernard, Paris
  - CHU Poitiers, Poitiers
  - Hôpital Pontchaillou, Rennes
  - CHU de Rouen, Rouen
  - Centre Cardiologique du Nord, Saint-Denis
  - CHU Strasbourg, Strasbourg
  - Clinique Pasteur, Toulouse
  - Hôpital Trousseau, Tours

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect the agreements made with funders.
  Teams wishing obtain IPD must meet the sponsor and PI team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasability and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).